CLINICAL TRIAL: NCT03333707
Title: Impact of a Mobile Application (Pacifica) on Stress, Anxiety, and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacifica Labs Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Pacifica Study 1
Record Dates: First submitted 2017-11-02; First posted 2017-11-07 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Anxiety; Stress; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Participants will be provided will full access to the Pacifica app.
  Interventions: Behavioral: Pacifica App
- Wait List (No Intervention): Participants will be placed on a wait list and will receive access to the app after 1 month.

INTERVENTIONS:
Behavioral: Pacifica App — The app contains several activities which are digital implementations of standard psychotherapy practices. Users may select which app elements they would like to use, and when. These app elements include relaxation and meditation activities, tools to examine your thoughts or self-talk, goal setting lists, and mood and health ratings. The app also has a peer support community where users can communicate with others who are having similar experiences. There is no minimum requirement for amount of time spent on any given activity, or in the app in total. The commercially available app has a feature to connect users to their existing healthcare providers, but this feature will not be available to study participants. Study participants may continue to see their existing providers.
  Arms: Active

SUMMARY:
The study is designed to examine the efficacy of a mobile application implementation of existing best practices in mental health treatment for managing stress, anxiety, and depression.

DETAILED DESCRIPTION:
Over 61 million adults in the U.S. experience mental illness in a given year, and only 1 in 3 will receive professional care due to difficulties with access to care, stigma, cost, or time involved in seeking treatment. Pacifica Labs, Inc., produces a Mobile Application ("app") which integrates existing best practices in treatment for stress, anxiety, and depression. One major goal of the app is to empower individuals to effectively self-manage their anxiety and depression. Pacifica has been used in a pilot research study, amongst a group of nonclinical college student volunteers. It was found to have a preventative effect on stress levels (as measured by the DASS-21). The current study is designed to consider a broader population of potential users.

Study Product Pacifica is a mobile app designed to teach users strategies to manage their stress, anxiety, and depression. Users can choose which tools they want to use. The strategies are digital implementations of existing practices in psychology such as thought records, mindfulness meditation & relaxation exercises, and behavioral activation. Pacifica includes optional "guided paths" of daily psychoeducation and and activities, which users can follow if they like. The app also includes features like mood and health tracking to help individuals notice patterns in their moods and make adjustments to their activities to manage their emotions more effectively. Additionally, there is a "hope board" which serves as a place for users to put inspirational quotes, reassuring photos, or save their completed activities to be reminded of their successes in using the app. Finally, the app offers a peer support community, which is a discussion board for users to connect with others going through similar experiences or who share interests.

The interventions based on Cognitive-Behavioral Therapy (CBT) include the "Thoughts" tool, which educates users about the effect of thinking errors or "cognitive distortions" on emotions and then prompts users to complete a text-based thought record, identify any cognitive distortions, and then challenge those thoughts (via positive reframe). The "Goals" tool is also based on CBT and allows users to create a list of goals to face their fears (in the case of anxiety) or re-engage with life (for those struggling with depression). The tool helps users to track their tasks and progress.

The interventions based on Mindfulness include "Meditations" which provides a suite of activities for users to learn mindfulness, practice deep breathing or body scans, guided relaxation activities, or simply listen to soothing sounds.

Pacifica also offers health-behavior tracking which allows users to monitor activities of their choice such as caffeine consumption, exercise, time spent with loved ones, etc. Users can also track their mood state "How are you feeling?" (scale of 1 = awful to 7 = great). Additionally, users can create and track custom health activities and associate words with their mood from pre-set options such as "stressed" or "happy" or can specify their own words using a hashtag such as "#engaged".

Users are able to see a visual display of their within-app self-monitoring data through the "Progress" function of the app.

The commercially available Pacifica app also allows users to connect to their health care providers through the "My Therapist" tab. This feature will be disabled for the present research study.

Participants in the study will be allowed to use whichever tools they want, in the same way that regular app users can. There is no minimum or maximum "dose" specified.

ELIGIBILITY:
Inclusion Criteria:

* Target disease: participants who score between 5 and 14 on the GAD-7 OR between 5 and 14 on the PHQ-8 and are therefore believed to be experience mild to moderate depression or anxiety
* No previous experience using the Pacifica app.
* Regular access to a smartphone
* Fluent in English
* Living in U.S.

Exclusion Criteria:

* Below 5 or over 14 on GAD-7 or below 5 or over 14 on PHQ-8
* Positive response on screener of presence of diagnosis of bipolar disorder, schizophrenia, other psychotic spectrum disorder, organic brain disease, currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Change in Depression | 2 weeks, 1 month, 3 months
  Change in Patient Health Questionnaire-8 (PHQ-8) score. Range is 0-24. Lower scores indicate less depression.
Change in Anxiety | 2 weeks, 1 month, 3 months
  Change in Generalized Anxiety Disorder-7 (GAD-7) score. Range is 0-19. Lower scores indicate less anxiety.
Change in Depression, Anxiety, Stress | 2 weeks, 1 month, 3 months
  Change in Depression Anxiety Stress Scale-21 (DASS-21) score. We will look at subscales. Ranges for depression, anxiety, and stress are 0-28, 0-20, and 0-33, respectively. Lower scores indicate less severity.

SECONDARY OUTCOMES:
Change in Self-Efficacy | 2 weeks, 1 month, 3 months
  Change in Score on General Self Efficacy Scale. Range is 10-40. Higher scores correspond to higher self-efficacy beliefs.

CONTACTS AND LOCATIONS:
Locations (1):
- Pacifica Labs, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not shared.

REFERENCES:
- [Derived] Moberg C, Niles A, Beermann D. Guided Self-Help Works: Randomized Waitlist Controlled Trial of Pacifica, a Mobile App Integrating Cognitive Behavioral Therapy and Mindfulness for Stress, Anxiety, and Depression. J Med Internet Res. 2019 Jun 8;21(6):e12556. doi: 10.2196/12556. PMID 31199319